CLINICAL TRIAL: NCT01280435
Title: Islide-Establishing a Clinical Dermatopathology Online Discourse System
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Yu-Chuan Li, Graduate Institute of Biomedical Informatics, Taipei Medical University
Other Study IDs: 99046
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Biopsy
Keywords: Online Discourse; e-Learning; Biopsy; Virtual Pathologic Section

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The trend is changed by a large number of low-cost computers, large-capacity computing power, and the rapid advent of network bandwidth. From the Internet to the WWW to Web2.0, the technology in addition brings impact on economic, social, and technological, but also on medical education about knowledge delivery globally and learning patterns.

Currently, many scholars start to take the affection of social network seriously. In the medical field, ECGpedia is the typical successful example. There are more than 250,000 members from 188 different countries in the website. On the other hand, the effect of data computing and transition improve the development of Gigapixel image presentation. For example, users can zoom in and zoom out on GoogleMap. The research team has being worked on this kind of search engine on pathology and anatomy slides in past three years. For education purpose, students can observe slides by using a virtual microscope directly.

This research will target on establishing a Clinical Dermatopathology Online Discourse System (iSlide). It will combine a virtual microscope platform and a biopsy diagnosis eLearning System. This survey will be focused on evaluating of this platform. The object is all interns in dermatopathology department at Wan Fang Hospital this semester. All the new physicians can learn from experienced experts. Users who have questions can search for help from others via this website. They can get assistance by thinking procedure learning model -scheme inductive and pattern recognition. In doing so, clinicians and pathologists can discuss with each other through this system. It also can improve the education and research development in this field.

ELIGIBILITY:
Inclusion Criteria:

* All interns in dermatology department of Wan Fang Hospital this semester.

Exclusion Criteria:

* N/A

Min Age: 20 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: interns
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-08; Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chuan Li, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan